CLINICAL TRIAL: NCT00110812
Title: STALWART: A Randomized, Open-Label, International Study of Subcutaneous Recombinant Interleukin-2 With and Without Concomitant Antiretroviral Therapy in Patients With HIV-1 Infection and CD4+ Cell Counts of 300 Cells/mm3 or More
Brief Title: Effect of Intermittent Aldesleukin Treatment With or Without Anti-HIV Drugs in HIV Infected People
Acronym: STALWART
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Chiron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ESPRIT 002; 10053 (Registry Identifier: DAIDS ES Registry Number); NCT00106730 (obsolete NCT alias)
Record Dates: First submitted 2005-05-13; First posted 2005-05-16 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2014-04

CONDITIONS: HIV Infections
Keywords: Treatment Naive; IL-2; rIL-2
MeSH Terms: conditions — HIV Infections | interventions — Interleukin-2; aldesleukin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- No IL-2 (No Intervention): Participants will receive no aldesleukin or HAART
- IL-2 without ART (Experimental): Participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level. Some Group 2 participants may take part in additional cycles of aldesleukin if they meet certain study criteria.
  Interventions: Drug: IL-2
- IL-2 with pericycle HAART (Experimental): Participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level; Group 3 participants will also take HAART for 3 days prior to the start of each aldesleukin cycle, throughout the 5-day aldesleukin cycle, and for 2 days after the end of each aldesleukin cycle (for a maximum of 10 days with each aldesleukin cycle). Some Group 3 participants may take part in additional cycles of aldesleukin if they meet certain study criteria. HAART is not supplied by the study, and choice of drugs is left to the participant and physician. The HAART regimen should include at least one protease inhibitor and at least 2 nucleoside/nucleotide reverse transcriptase inhibitors.
  Interventions: Drug: IL-2

INTERVENTIONS:
Drug: IL-2 — 7.5 MIU injected intramuscularly; one arm uses Proleukin together with HAART of choice (protease inhibitor and at least 2 nucleoside/nucleotide reverse transcriptase inhibitors)
  Other Names: Proleukin, Aldeskeukin
  Arms: IL-2 with pericycle HAART; IL-2 without ART

SUMMARY:
The purpose of this study is to determine the effect of short cycles of recombinant interleukin-2 (also known as rIL-2 or aldesleukin) given with or without anti-HIV drugs in HIV infected patients. The effects will be compared with a study group that receives no IL-2 or antiretroviral therapy.

Study hypothesis: Intermittent aldesleukin, when given without antiretroviral therapy to patients with early HIV infection, will produce no change in HIV viral load and increases in CD4+ T lymphocyte counts comparable to aldesleukin administered with antiretrovirals.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) has dramatically improved prognosis and lowered morbidity and mortality rates for HIV infected patients. However, significant drug toxicities, difficulties with patient compliance to HAART regimens, and development of drug resistance highlight the need for less toxic, immune-based strategies. Aldesleukin is a synthetic protein that can increase CD4 counts; it is currently approved by the Food and Drug Administration (FDA) for use in patients with metastatic melanoma and renal cell carcinoma. Previous studies of aldesleukin in HIV infected patients indicated that increased CD4 counts can persist for years after aldesleukin administration, and aldesleukin given with HAART may also lead to significant lowering of viral load. This study will examine the immunologic effects of intermittent cycles of aldesleukin administered with and without HAART as compared to no therapy in HIV infected patients.

This study will last approximately 31 months. Participants will be randomly assigned to one of three groups at study entry. Group A will receive no aldesleukin or HAART. Group B will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level. Group C will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level; Group C participants will also take HAART for 3 days prior to the start of each aldesleukin cycle, throughout the 5-day aldesleukin cycle, and for 2 days after the end of each aldesleukin cycle (for a maximum of 10 days with each aldesleukin cycle). HAART will not be provided by the study. Some Group B and C participants may take part in additional cycles of aldesleukin if they meet certain study criteria.

All participants in this study will have at least 8 study visits; these visits will occur at study entry and Weeks 4, 8, 12, 16, 20, 24, and 32. Blood collection will occur at all visits and will include tests for CD4 count and viral load. Groups B and C will have additional blood collection within 4 days prior to the start of each aldesleukin cycle. On the last day of each aldesleukin cycle, Groups B and C will be assessed for toxicities, adverse events, and adherence to the aldesleukin daily injections; they will also have another blood collection. Group C participants will have an additional blood collection for HIV genotyping after they have completed their third aldesleukin cycle. Extended follow-up visits will occur approximately every 4 months for an additional two years. Blood collection will occur at these visits and will include tests for CD4 count, viral load, and other laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* HIV infected
* CD4 count of 300 cells/mm3 or more
* Access to a HAART regimen consisting of 1 or more protease inhibitors (PIs) and 2 or more nucleoside or nucleotide reverse transcriptase inhibitors

Exclusion Criteria:

* Prior use of aldesleukin
* Approved or experimental antiretroviral drug (including hydroxyurea) within 1 year prior to study entry
* Evidence of virologic failure on a PI- or nonnucleoside-based HAART regimen
* Any current indication for continuous HAART, in the opinion of the investigator
* Any contraindication to HAART, in the opinion of the investigator
* Systemic corticosteroids, chemotherapy, or experimental cytotoxic drugs within 45 days of randomization
* Approved or experimental agents with clinically significant immunomodulatory effects within 8 weeks prior to randomization
* History of any AIDS-defining illness or certain other diseases. More information on this criterion can be found in the protocol.
* Concurrent cancer requiring cytotoxic therapy
* Any central nervous system (CNS) abnormality requiring ongoing treatment with antiseizure medication
* Current or prior autoimmune or inflammatory diseases, including inflammatory bowel disease, psoriasis, optic neuritis, or any other autoimmune or inflammatory diseases with potentially life-threatening complications
* Significant heart, lung, kidney, liver, gastrointestinal, CNS, or psychiatric disease OR illicit substance use or abuse that, in the opinion of the investigator, would interfere with the study
* Pregnancy or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 267 (Actual)
Dates: Start 2005-09; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jorge Tavel, MD, Study Chair — National Institute for Allergy and Infectious Diseases, National Institutes of Health
Locations (36):
- United States (11):
  - VA Greater Los Angeles Healthcare System, Infectious Diseases Section CRS, Los Angeles, California
  - Washington DC VAMC, Washington Regional AIDS Program, Infectious Diseases CRS, Washington D.C., District of Columbia
  - NIH Clinical Ctr., NIAID HIV Clinic CRS, Bethesda, Maryland
  - Henry Ford Hosp. CRS, Detroit, Michigan
  - Harlem Hospital Ctr./Columbia University CRS (Gordin CTU), New York, New York
  - Lincoln Hosp. & Med. Ctr. CRS, The Bronx, New York
  - Providence Portland Med. Ctr., Ambulatory Care and Education Ctr. CRS, Portland, Oregon
  - Michael E. DeBakey VAMC CRS, Houston, Texas
  - Thomas Street Clinic CRS, Houston, Texas
  - South Texas Veterans Health Care System, Immunosuppression Clinic CRS, San Antonio, Texas
  - Virginia Commonwealth Univ. Medical Ctr. CRS, Richmond, Virginia
- Argentina (4):
  - Hosp. Italiano de Buenos Aires, Infectious Diseases Section CRS, Ciudad de Buenos Aires, Buenos Aires
  - Hosp. Gen. de Agudos JM Ramos Mejia, Servicio de Inmunocomprometidos CRS, Ciudad de Buenos Aires, Buenos Aires
  - Funcei Crs, Ciudad de Buenos Aires, Buenos Aires
  - Caici Crs, Rosario, Provincia de Sante Fe
- Australia (5):
  - St. Vincent's Hospital CRS, Darlinghurst, New South Wales
  - Queensland Health - AIDS Med. Unit CRS, Brisbane, Queensland
  - Gladstone Road Medical Ctr. CRS, Highgate Hill, Queensland
  - Gold Coast Sexual Health Clinic CRS, Miami, Queensland
  - Carlton Clinic CRS, Carlton, Victoria
- Fundacion Arriaran CRS, Santiago, Chile
- Italy (2):
  - Ospedale San Raffaele S.r.l. CRS, Milan
  - Univ. of Milan, Ospedale Luigi Sacco, Institute of Infectious and Tropical Diseases CRS, Milan
- Univ. Hosp. Ctr. of the Med. School of Casablanca, Infectious Diseases Unit CRS, Casablanca, Morocco
- Wojewodzki Szpital Zakazny CRS, Warsaw, Poland
- Portugal (3):
  - Hospital de Cascais, HDDI, Departamento Medicina Interna CRS, Cascais
  - Hosp. de Egas Moniz, Servicio de Infecciologia e Medicina Tropical CRS, Lisbon
  - Hosp. de Santa Maria, Servico de Doencas Infecciosas CRS, Lisbon
- Hosp. Clinico de Barcelona CRS, Barcelona, Spain
- Thailand (3):
  - Chulalongkorn University Hospital CRS, Bangkok, Ratchathewi
  - Chiang Rai Regional Hosp. INSIGHT CRS, Chiangrai
  - Khon Kaen Univ., Srinagarind Hosp., Div. of Infectious Diseases & Tropical Medicine, Dept. of Medici, Khon Kaen
- United Kingdom (4):
  - Brighton & Sussex Univ. Hosp. NHS Trust, HIV Research Office CRS, Elm Grove, Brighton
  - Leicester Royal Infirmary, Dept. of Infection & Tropical Medicine CRS, Leicester
  - St. Bartholomew's Hosp., Infection & Immunity Clinical Group CRS, London
  - St. Mary's Hosp. of London, Imperial College School of Medicine CRS, London

REFERENCES:
- [Background] Anaya JP, Sias JJ. The use of interleukin-2 in human immunodeficiency virus infection. Pharmacotherapy. 2005 Jan;25(1):86-95. doi: 10.1592/phco.25.1.86.55629. PMID 15767224
- [Background] de Boer AW, Markowitz N, Lane HC, Saravolatz LD, Koletar SL, Donabedian H, Yoshizawa C, Duliege AM, Fyfe G, Mitsuyasu RT. A randomized controlled trial evaluating the efficacy and safety of intermittent 3-, 4-, and 5-day cycles of intravenous recombinant human interleukin-2 combined with antiretroviral therapy (ART) versus ART alone in HIV-seropositive patients with 100-300 CD4+ T cells. Clin Immunol. 2003 Mar;106(3):188-96. doi: 10.1016/s1521-6616(02)00038-4. PMID 12706405
- [Background] Davey RT Jr, Murphy RL, Graziano FM, Boswell SL, Pavia AT, Cancio M, Nadler JP, Chaitt DG, Dewar RL, Sahner DK, Duliege AM, Capra WB, Leong WP, Giedlin MA, Lane HC, Kahn JO. Immunologic and virologic effects of subcutaneous interleukin 2 in combination with antiretroviral therapy: A randomized controlled trial. JAMA. 2000 Jul 12;284(2):183-9. doi: 10.1001/jama.284.2.183. PMID 10889591
- [Background] Marchetti G, Franzetti F, Gori A. Partial immune reconstitution following highly active antiretroviral therapy: can adjuvant interleukin-2 fill the gap? J Antimicrob Chemother. 2005 Apr;55(4):401-9. doi: 10.1093/jac/dkh557. Epub 2005 Feb 24. PMID 15731201
- [Background] Pett SL, Kelleher AD. Cytokine therapies in HIV-1 infection: present and future. Expert Rev Anti Infect Ther. 2003 Jun;1(1):83-96. doi: 10.1586/14787210.1.1.83. PMID 15482104
- [Derived] Tavel JA; INSIGHT STALWART Study Group; Babiker A, Fox L, Gey D, Lopardo G, Markowitz N, Paton N, Wentworth D, Wyman N. Effects of intermittent IL-2 alone or with peri-cycle antiretroviral therapy in early HIV infection: the STALWART study. PLoS One. 2010 Feb 23;5(2):e9334. doi: 10.1371/journal.pone.0009334. PMID 20186278

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled by HIV care providers between December 2005 and June 2008. When the main study ended in February 2009, patients who consented to a study extension were followed another 2 years, during which study drug was not given.
Groups:
- No IL-2: Participants will receive no aldesleukin or HAART during the main study or extension
- IL-2 Without ART: During the main study, participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level. Patients did not receive aldesleukin during the extension phase.
- IL-2 With Pericycle HAART: During the main study, participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level; in addition, this group will also take HAART for 3 days prior to the start of each aldesleukin cycle, throughout the 5-day aldesleukin cycle, and for 2 days after the end of each aldesleukin cycle (for a maximum of 10 days with each aldesleukin cycle). Patients did not receive aldesleukin during the extension phase.
Period: Main Study
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Started | 91 | 89 | 87
Completed | 83 | 78 | 74
Not Completed | 8 | 11 | 13
Not completed — Death | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 1
Not completed — Lost to Follow-up | 8 | 11 | 10
Period: Extended Follow-up
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Started | 80 | 69 | 73
Completed | 78 | 65 | 69
Not Completed | 2 | 4 | 4
Not completed — Death | 1 | 0 | 3
Not completed — Withdrawal by Subject | 0 | 1 | 0
Not completed — Lost to Follow-up | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- IL-2 Without ART: Participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level.
- IL-2 With Pericycle HAART: Participants will receive aldesleukin under the skin twice daily for 5 consecutive days every 8 weeks for 3 cycles, then as needed to maintain CD4 counts at or above a goal level; in addition, this group will also take HAART for 3 days prior to the start of each aldesleukin cycle, throughout the 5-day aldesleukin cycle, and for 2 days after the end of each aldesleukin cycle (for a maximum of 10 days with each aldesleukin cycle).
- Total: Total of all reporting groups
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART | Total
Number analyzed (Participants) | 91 | 89 | 87 | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 91 | 89 | 85 | 265
  >=65 years | 0 | 0 | 2 | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.1 (7.7) | 37.3 (9.6) | 37.8 (11.0) | 37.4 (9.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 17 | 13 | 46
  Male | 75 | 72 | 74 | 221
Region of Enrollment [Number; unit: participants]
  Portugal | 3 | 3 | 4 | 10
  United States | 8 | 9 | 9 | 26
  Morocco | 1 | 0 | 0 | 1
  Argentina | 25 | 24 | 21 | 70
  Thailand | 21 | 21 | 22 | 64
  Spain | 1 | 1 | 1 | 3
  Poland | 3 | 2 | 3 | 8
  Australia | 10 | 8 | 8 | 26
  Chile | 2 | 5 | 4 | 11
  United Kingdom | 8 | 9 | 10 | 27
  Italy | 9 | 7 | 5 | 21
CD4 cell count [Median (Inter-Quartile Range); unit: cells/mm^3] | 432 [375 to 507] | 398 [355 to 458] | 425 [365 to 535] | 418 [359 to 511]

OUTCOME MEASURES:

1. Primary Outcome: Mean Change in CD4+ T Lymphocyte Count
Description: Change in CD4 count from baseline to week 32.
Time Frame: Week 32
Population: patients for whom the week-32 CD4+ cell count was measured
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 83 | 78 | 74
cell/mm^3 | -21.8 (93.1) | 113.7 (216.8) | 110.4 (174.7)
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p < .001, ANOVA — Adjusted for 3 pairwise comparisons; stratified by geographic region and adjusted for baseline CD4; Mean Difference (Net) = 134, 95% CI 2-sided [70 to 198]
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p < .001, ANOVA — Adjusted for 3 pairwise comparisons; stratified by geographic region and adjusted for baseline CD4; Mean Difference (Net) = 133, 95% CI 2-sided [68 to 199]

2. Secondary Outcome: Discontinuation of IL-2
Description: Patients receiving fewer than 3 cycles of IL-2 by week 32
Time Frame: week 32
Population: all patients randomized to a study arm containing IL-2
Measure: Number; unit: participants
Arm/Group | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 89 | 87
participants | 12 | 32

3. Secondary Outcome: Plasma HIV RNA
Description: change from baseline in HIV-RNA copies/ml (log10)
Time Frame: At Week 32
Population: Patients for whom HIV-RNA was available at week 32
Measure: Mean (Standard Deviation); unit: copies/ml (log 10)
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 82 | 79 | 72
copies/ml (log 10) | -.39 (1.03) | -.07 (.80) | -.01 (.40)
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p = .01, ANOVA; stratified by region and adjusted for baseline HIV-RNA; Mean Difference (Net) = .31, 95% CI 2-sided [.08 to .54]
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p = .003, ANOVA; stratified by region and adjusted for baseline HIV-RNA; Mean Difference (Net) = .36, 95% CI 2-sided [.12 to .60]

4. Secondary Outcome: Change in CD4 T Lymphocyte Count
Description: change from baseline to month 12 in CD4 T lymphocyte count
Time Frame: At Month 12
Population: patients for whom the month 12 CD4 count was available
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 78 | 77 | 72
cell/mm^3 | -8.4 (129.1) [356 to 472] | 59.0 (176.0) [357 to 589] | 49.8 (155.6) [359 to 605]
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p = .009, ANOVA; ANOVA with stratification by region and adjustment for baseline CD4; Mean Difference (Net) = 65.8
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p = .02, ANOVA; stratified by region and adjusted for baseline CD4; Mean Difference (Net) = 58.2

5. Secondary Outcome: HIV-1 Genotype Changes
Description: Patients who developed mutations associated with antiretroviral drugs.
Time Frame: after 3rd cycle of IL-2
Population: Per protocol, the analysis of genotypic changes associated with antiretroviral resistance was restricted patients in one arm, namely, patients assigned to take pericycle HAART who completed 3 cycles of IL-2 and who had successful genotypes.
Measure: Number; unit: participants
Arm/Group | IL-2 With Pericycle HAART
Number analyzed (Participants) | 47
participants | 2

6. Secondary Outcome: Fasting Lipid Profile
Description: total fasting cholesterol
Time Frame: week 32
Population: all patients with laboratory data at week 32 who reported fasting
Measure: Mean (Standard Deviation); unit: mg/dl
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 65 | 66 | 58
mg/dl | 173.4 (33.7) | 167.0 (32.7) | 164.6 (40.8)

7. Secondary Outcome: Disease Progression or Death
Description: occurrence of an opportunistic event (AIDS-defining infection or malignancy) or death
Time Frame: throughout study, through Feb 28 2009 (median followup of 19 months)
Population: all randomized patients
Measure: Number; unit: participants
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 91 | 89 | 87
participants | 1 | 5 | 7
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p = .14, Regression, Cox; Unadjusted, stratified by region; Hazard Ratio (HR) = 5.08, 95% CI 2-sided [0.59 to 43.6] — Patients taking IL-2 alone compared to patients not taking IL-2
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p = .08, Regression, Cox; Unadjusted, stratified by region; Hazard Ratio (HR) = 6.56, 95% CI 2-sided [0.80 to 53.6] — Patients taking IL-2 plus pericycle HAART compared to patients not receiving IL-2

8. Secondary Outcome: Initiation of Continuous ART
Description: While patients were not taking ART at baseline or while undergoing IL-2 cycles (other than use of pericycle ART in one of the three groups), some chose to start an ART regimen during the study.
Time Frame: from randomization through February 28, 2009
Population: all patients randomized
Measure: Number; unit: participants
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 91 | 89 | 87
participants | 34 | 23 | 14
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p = .048, Regression, Cox; Hazard Ratio (HR) = .58, 95% CI 2-sided [.34 to .99] — IL-2 without ART vs control group
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p < .001, Regression, Cox; Hazard Ratio (HR) = .32, 95% CI 2-sided [.17 to .62] — IL-2 with pericycle HAART compared to control

9. Secondary Outcome: Change in HIV-RNA Copies/ml (log10) From Baseline to Month 12
Time Frame: month 12
Population: patients for whom HIV-RNA measurement was available at baseline and month 12.
Measure: Mean (Standard Deviation); unit: copies/ml (log 10)
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 77 | 74 | 71
copies/ml (log 10) | -0.64 (1.24) [1740 to 25771] | -0.28 (0.95) [1794 to 69953] | -0.09 (0.84) [7790 to 49183]
Statistical Analysis 1: Comparison: No IL-2 vs IL-2 Without ART; Test type: Superiority or Other; p = .03, ANOVA; Stratified by region and adjusted for baseline HIV-RNA; Mean Difference (Net) = 0.34, 95% CI 2-sided [0.03 to 0.64]
Statistical Analysis 2: Comparison: No IL-2 vs IL-2 With Pericycle HAART; Test type: Superiority or Other; p < .001, ANOVA; Stratified by region and adjusted for baseline HIV-RNA; Mean Difference (Net) = 0.54, 95% CI 2-sided [0.24 to 0.85]

10. Secondary Outcome: Thyroid Stimulating Hormone
Description: Number of participants with thyroid stimulating hormone greater than the upper limit of normal
Time Frame: week 32
Population: all patients with TSH measured at 32 weeks
Measure: Number; unit: participants
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 79 | 75 | 71
participants | 3 | 2 | 7

11. Secondary Outcome: SGOT
Description: Number of participants with aspartate aminotransferase (SGOT) greater than 5 times the upper limit of normal
Time Frame: week 32
Population: all patients with SGOT measured at week 32
Measure: Number; unit: participants
Arm/Group | No IL-2 | IL-2 Without ART | IL-2 With Pericycle HAART
Number analyzed (Participants) | 83 | 79 | 74
participants | 1 | 0 | 0

12. Post Hoc Outcome: Opportunistic Disease or Death During the Trial Extension Phase
Description: Incidence of an opportunistic event (AIDS-defining infection or malignancy) or death between February 28, 2009, when the main study ended, and February 28, 2011, when the extended phase was completed.
Time Frame: two years following close of main study
Population: All patients who were alive at the end of the main study and who consented to be followed for an additional 2 years in the extension phase. Because the focus of the extension was on the safety of patients exposed to IL-2, the outcomes were summarized for the two groups exposed to IL-2 vs. the group that did not take IL-2.
Measure: Number; unit: participants
Groups:
- IL-2: Consenting patients who were assigned IL-2 during the main phase of the study, including patients who took IL-2 alone as well as patients who took IL-2 with ART.
- Control: Consenting patients who were in the control group during the main phase of the trial.
Arm/Group | IL-2 | Control
Number analyzed (Participants) | 142 | 80
participants | 8 | 3
Statistical Analysis 1: Comparison: IL-2 vs Control; Test type: Superiority or Other; p = .59, Regression, Cox; Stratification by region; Hazard Ratio (HR) = 1.45, 95% CI 2-sided [0.38 to 5.45] — IL-2 group compared to control group

13. Post Hoc Outcome: CD4+ Cell Count 2 Years Post-study
Time Frame: two years following close of main study
Population: All patients for whom a CD4 count measurement was available during the extension phase. Because the focus of the extension was on the safety of patients exposed to IL-2, the outcomes were summarized for the two groups exposed to IL-2 vs. the group that did not take IL-2.
Measure: Mean (Standard Deviation); unit: cell/mm^3
Arm/Group | IL-2 | Control
Number analyzed (Participants) | 141 | 80
cell/mm^3 | 499.9 (191.4) | 557.2 (225.5)
Statistical Analysis 1: Comparison: IL-2 vs Control; Test type: Superiority or Other; p = .05, ANOVA; Last measured CD4 is imputed if month 24 CD4 count is missing. Analysis is adjusted for baseline CD4; Mean Difference (Final Values) = -55.9, Standard Error of Mean 28.4 — IL-2 group minus control group CD4

14. Post Hoc Outcome: Undetectable HIV-RNA
Description: Patients with undetectable HIV-RNA levels measured at 24 months after the close of the main study, at the end of the extension phase.
Time Frame: 24 months post-trial
Population: All patients for whom an HIV-RNA measurement was available during the extension phase. Because the focus of the extension was on the safety of patients exposed to IL-2, the outcomes were summarized for the two groups exposed to IL-2 vs. the group that did not take IL-2.
Measure: Number; unit: participants
Arm/Group | IL-2 | Control
Number analyzed (Participants) | 141 | 80
participants | 97 | 60

15. Post Hoc Outcome: Commencement of Continuous Antiretroviral Treatment
Description: Number of patients commencing continuous antiretroviral treatment.
Time Frame: from randomization through February 28, 2011, the end of the extension phase
Population: All randomized patients are counted. Patients who did not consent to the extension phase are censored at the end of the main study (Feb 28, 2009). Because the focus of the extension was on the safety of patients exposed to IL-2, the outcomes were summarized for the two groups exposed to IL-2 vs. the group that did not take IL-2.
Measure: Number; unit: participants
Arm/Group | IL-2 | Control
Number analyzed (Participants) | 176 | 91
participants | 108 | 66
Statistical Analysis 1: Comparison: IL-2 vs Control; Test type: Superiority or Other; p = .03, Regression, Cox; Hazard Ratio (HR) = .71, 95% CI 2-sided [.52 to .97] — IL-2 groups vs. control

ADVERSE EVENTS:
Time Frame: From randomization through Feb 28 2011, end of extended followup.
Description: Adverse events were recorded if grade 3 (moderate) or 4 (serious), according to DAIDS toxicity table.
Arm/Group | IL-2 With Pericylce HAART | IL-2 Without ART | No IL-2
Serious Adverse Events (participants affected / at risk) | 6/87 | 6/89 | 3/91
Other Adverse Events (participants affected / at risk) | 7/87 | 3/89 | 3/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-2 With Pericylce HAART (N=87) | IL-2 Without ART (N=89) | No IL-2 (N=91)
Anaemias NEC (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1)
Bacterial infections NEC (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Bladder and urethral symptoms (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Bronchospasm and obstruction (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Calcium metabolism disorders (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis and cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (excl infective) (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Ear infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Febrile disorders (General disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal atonic and hypomotility disorders NEC (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal and gastrointestinal infections (Infections and infestations) | 0 (0) | 0 (0) | 2 (2)
General nutritional disorders NEC (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Hyperparathyroid disorders (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0)
Non-site specific injuries NEC (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Renal failure and impairment (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Male reproductive tract infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Salivary gland disorders NEC (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Central nervous sytem haemorrhages and cerebrovascular accidents (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Chemical injuries (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disorders NEC (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Depressive disorders (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2)
Epstein-Barr viral infections (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pulmonary thrombotic and embolic conditions (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Sepsis, bacteraemia, viraemia and fungaemia NEC (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | IL-2 With Pericylce HAART (N=87) | IL-2 Without ART (N=89) | No IL-2 (N=91)
Febrile disorders (General disorders) | 7 (7) | 3 (3) | 0 (0)
Abdominal and gastrointestinal infections (Infections and infestations) | 0 (0) | 0 (0) | 3 (3)

LIMITATIONS AND CAVEATS:
All randomized patients were followed through 28 Feb 2009. A subset of 222 consenting patients were followed 2 additional years, through 28 Feb 2011.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes